CLINICAL TRIAL: NCT04779762
Title: Stelara and CDED Diet Trial for Crohn"s Disease
Brief Title: Stelara and Diet Trial for Crohn"s Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Wolfson Medical Center (Other Government)
Collaborators: Sheba Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STEDI
Record Dates: First submitted 2021-02-28; First posted 2021-03-03 (Actual); Last update posted 2021-03-03 (Actual); Status verified 2021-02

CONDITIONS: Crohn Disease
MeSH Terms: conditions — Crohn Disease | interventions — Ustekinumab

STUDY DESIGN:
Who Masked: Investigator
Masking Description: single blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental): Standard induction regimen of Ustekinumab with the Crohn's disease exclusion diet (CDED)
  Interventions: Other: Crohn's disease exclusion diet (CDED); Drug: Ustekinumab Injection [Stelara]
- Group 2 (Active Comparator): Standard induction regimen of Ustekinumab as above without diet
  Interventions: Drug: Ustekinumab Injection [Stelara]

INTERVENTIONS:
Other: Crohn's disease exclusion diet (CDED) — Dietary therapy for Crohn's disease
  Arms: Group 1
Drug: Ustekinumab Injection [Stelara] — Drug for Crohn's disease

SUMMARY:
Dietary therapy involving the Crohn's disease exclusion diet (CDED) is an evolving strategy to target the microbiome and innate immunity in order to reduce inflammation and promote healing.

The goal of the current pilot study is to evaluate the added benefit of treatment with Ustekinumab combined with CDED in anti TNF exposed patients compared to treatment with Ustekinumab alone in term of achieving remission.

DETAILED DESCRIPTION:
The induction period is crucial for a patient's response to biologic therapy but also for maintenance of remission, as simple as it sounds, maintenance of remission requires remission. Biological medications using a single monoclonal antibody directed target, seem to be effective only for a segment of the population with Crohn's disease Dietary therapy is highly effective in children and induces remission in approximately 60% of young adults with uncomplicated luminal disease. It was shown to shift the microbiome away from Proteobacteria towards Firmicutes, and to decrease intestinal permeability (i.e improvement in leaky gut).

Dietary therapy is widely used in children and both exclusive enteral nutrition (EEN) and the Crohn's disease exclusion diet were highly effective for induction of remission and reduction in inflammation in children in a multinational randomized controlled trial (Levine A, Gastroenterology 2019). Recently a prospective randomized controlled trial in biologic naïve adults demonstrated clinical remission in 62% of adults by 6 weeks (Yanai H, UEG Week 2020). A two week course of EEN in adults was effective for improvement of symptoms and reduction in inflammation (Wall CL Inflamm Intest Dis 2018). Xu et al demonstrated clinical remission in 52 and 47% of two adult cohorts (n=104) using EEN for induction of remission (Xu Y, Therap Adv Gastroenterol 2019). Taken together, these studies suggest that dietary therapy could act as a bridge to biologic effect and have a synergistic effect on the disease.

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent.
2. Age: 18- 65 years (inclusive).
3. Established diagnosis of CD
4. Starting Ustekinumab.
5. Active disease defined as a CDAI >220, and have an objective measure of disease activity such as an elevated marker of inflammation (elevated CRP >5mg/L or 0.5 mg/dL or calprotectin >150 mcg/g).
6. Patients must have previously received at least one dose of anti TNF at any time in the past.
7. Stable medication at least 8 weeks.

Inclusion criteria comments

1. Patients of any weight will be recruited and randomized to the study regardless of their BMI.

Exclusion Criteria:

1. Pregnancy or lactation
2. Presence of malignancy
3. Use of prednisone >20 mg /day
4. Ongoing use of concurrent medications with a dose change in the previous 8 weeks with the exception of steroids (Patients receiving prednisone 20 mg or less may be enrolled by must be tapered by week 6).
5. Treatment with an anti TNF in the last 4 weeks.
6. Patients who will take oral iron oral supplements during the trial (see comment 1 below).
7. Active infections, tuberculosis, positive stool test for Clostridium difficile toxin.
8. Active perianal fistula (with discharge, or with an abscess during the past 3 months), rectovaginal fistula.
9. Fever.
10. Active extra intestinal disease (arthritis with joint swelling, concurrent liver disease). Patients with skin manifestations and arthralgia may be included.
11. Smokers who smoke >5 more cigarettes a day (see comment 2 below).
12. Renal failure.
13. Uncontrolled diabetes that precludes the diet.
14. Patients with isolated colonic disease distal to the transverse colon (see comment 3 below).

Exclusion criteria comments

1. Patients taking oral iron supplements may be enrolled if they discontinue the supplements prior to receiving UST, and are NOT ALLOWED to take oral iron supplements during the first 12 weeks of the trial as the diet reduces oral iron exposure to decrease siderophoric pathobionts (patients are allowed to receive intravenous iron or other oral vitamins during the trial).
2. Patients who smoke >5 cigarettes per day may be enrolled if they stop smoking from the start of the trial (smoking negates the effect of the diet).
3. Patients with isolated colonic disease distal to the transverse colon and no history of ileal disease will be excluded to make sure that IBDU is not recruited.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-01 (Estimated); Primary Completion 2025-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
ITT, steroid free remission | week 12
  Defined as an improvement in one inflammatory marker (CRP or calprotectin)

SECONDARY OUTCOMES:
Median calprotectin | week 12
  Reduction in median calprotectin compared to baseline between groups
Intestinal bowel wall thickness | week 16
  Reduction in intestinal bowel wall thickness compared to baseline between groups for patients with increased bowel wall thickness measured on baseline US.
UST trough level | week 16
  mean UST trough level between groups.
CDAI between groups | week 16
  Median decline in CDAI between groups. Crohn's Disease Activity Index (CDAI) range between 0-800

CONTACTS AND LOCATIONS:
Locations (1):
- Sheba Medical Center, Ramat Gan, Israel

IPD SHARING:
Plan to Share IPD: Undecided